CLINICAL TRIAL: NCT05994300
Title: Clinical Research of Moderately Hypofractionated Radiotherapy for Cervical Cancer
Brief Title: Moderately Hypofractionated Adaptive Radiotherapy for Cervical Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHARTCC-Trial
Record Dates: First submitted 2023-08-05; First posted 2023-08-16 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Cervical Neoplasm; Adaptive Radiotherapy; Radiotherapy; Adverse Effect
Keywords: moderately hypofractionated radiotherapy; adaptive radiotherapy; cervical cancer.
MeSH Terms: conditions — Uterine Cervical Neoplasms; Radiation Injuries | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moderately Hypofractionated Adaptive Radiotherapy (Experimental)
  Interventions: Radiation: Moderately hypofractionated adaptive radiotherapy (ART)+ High-dose rate (HDR) Brachytherapy

INTERVENTIONS:
Radiation: Moderately hypofractionated adaptive radiotherapy (ART)+ High-dose rate (HDR) Brachytherapy — Experimental: 43.35Gy/17F external beam radiotherapy (EBRT) with adaptive radiotherapy (ART) + HDR-Brachytherapy
  Drug: Concurrent Chemotherapy
  Weekly cisplatin 40 mg/m2

SUMMARY:
External radiation given in 25 fractions or so together with weekly chemotherapy and followed by 5 or 6 fractions of brachytherapy is the standard of care for patients with locally advanced cervical cancer. We hope to develop external moderately hypofractionated radiotherapy of cervical cancer based on adaptive radiotherapy.The objective of this study is to evaluate the efficacy and treatment-related toxicity of moderately hypofractionated adaptive radiotherapy in the treatment of cervical cancer.

DETAILED DESCRIPTION:
This is an investigator-initiated efficacious, single-center, open-label clinical trial study. This study hypothesizes that the use of external moderately hypofractionated radiotherapy of cervical cancer based on adaptive radiotherapy. A dose of 43.35Gy in 17 fractions is delivered to clinical target volume (CTV). Patients receive cisplatin based concurrent chemotherapy. The primary endpoint is acute toxicity.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years to 70 years

FIGO Stage IB1, IB2, IB3, IIA or IIB cervical cancers

FIGO stage IIIC1 cervical cancers are candidates but must meet all the following criteria:largest node is less than 1.5 cm,less than 3 pathological nodes,No nodes located in the common iliac chain

Histology: squamous

Candidate for definitive chemoradiotherapy to be delivered with weekly cisplatin

Brachytherapy candidate

Functional State Eastern Cooperative Oncology Group (ECOG)0-2

Exclusion Criteria:

Patients who had chemotherapeutic, surgical and/or radiotherapy treatment

FIGO stage IIIA, IIIB, IIIC2, IVA or IVB

FIGO stage IIIC1 with node greater than 1.5 cm, common iliac node or greater than 2 pathological nodes

Previous pelvic or abdominal radiotherapy

Patient unable to undergo MR scan

ECOG performance status greater than 2

Not a cisplatin candidate

Other factors that contraindicate experimental therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 3 months
  This outcome is assessed by physicians during each follow-up appointment, and scored according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 . Clinically relevant toxicities of gastrointestinal, genitourinary, vaginal and non-specific general symptoms (i.e. fatigue, malaise and pain) will be collected. Hematological disorders will also be collected through weekly blood work checks. Acute toxicities will be collected at baseline, and then weekly during radiotherapy/chemoradiotherapy and at 3 months after completion of radiation.

SECONDARY OUTCOMES:
Late toxicity | 3 years
  Late toxicities will be collected from 3 months after completion of radiation onwards until the end of follow-up.
Response evaluation evaluated with RECIST 1.1 | One month after treatment
  Evaluated with RECIST 1.1
Disease-free survival | 3 years
  Disease-free survival was defined as the period from the diagnosis of cervical cancer to events that included death or disease progression at local, regional, or distant sites or until the date of the last follow-up.
Overall survival | 3 years
  Overall survival was defined as the period from the diagnosis of cervical cancer to the date of death or last follow-up.
Quality of life (QoL) | 3 years
  QoL will be measured by the cervical cancer module (QLQ-CX24). QLQ-CX24 includes cancer - and treatment - related items and symptoms regarding sexuality.
Quality of life (QoL) | 3 years
  QoL will evaluated by the EORTC QLQ-C-30 questionnaire.QLQ-C30 questionnaire is used for all cancers and has several symptom scales, five functional scales (physical, emotional, social, role, cognitive) and a global health status scale. Response options are a four-point Likert scale from "not at all" to "very much" or a seven-point Likert scale from "very poor" to "excellent."
Assessment of tumor regression throughout EBRT | 3 months
  To be assessed through volumetric comparison of tumor volume in the pre-EBRT and post-EBRT MRI scans.

CONTACTS AND LOCATIONS:
Overall Officials: Fuquan Zhang, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of the patients